Title: Development of innovative technologies for the treatment of pulmonary and heart failure to prolong human's life

NCT number: Will be provided

**Date:** 01.01.2021

#### 1. Annotation

There are used multiple techniques to reduce the syndrome of systemic inflammatory response, immunocorrection, and others in order to improve the results of implantation of mechanical devices, patients on the extracorporeal life-sustaining system and septic patients before surgery. Today, there are many ways to prevent the development of a systemic inflammatory response by removing leukocytes from the bloodstream by integrating a filter with a special screen in the perfusion circuit to remove leukocytes and prevent the latter from entering the systemic circulation.

The most effective approach is the method of extracorporeal hemadsorption, intended for additional therapy of patients with an increased level of cytokines in conditions of the systemic inflammatory response syndrome, in which a patient with acute pulmonary distress syndrome and cardiogenic septic shock against the background of an extracorporeal hemofiltration, an extracorporeal cytokine adsorber system was installed, intended to eliminate a wide range of inflammatory mediators, as well as multiple proteins and metabolites.

# The purpose of the program.

Formulation of new treatments for heart and pulmonary failure through using organreplacing technologies.

Formulation of a clinical protocol and implementation of treatment methods into clinical practice heart and pulmonary failure using organ-replacing technologies.

## Study design.

Study type: interventional (clinical study)

Set of participants: 100 participants

Distribution: randomized

Interventional model: parallel

Masking: no

.14.011111.8. 110

Primary Goal: Treatment

New methods were created for rehabilitating the function of affected organs after implantation of the LVAD, a total artificial heart, an extracorporeal life-sustaining system will be of great importance, both for Kazakhstan and for states with similar problems of donor organ deficiency, will also improve the effectiveness of surgical treatment and reduce

the level of complications and mortality of patients on the extracorporeal life-sustaining system and septic patients.

Furthermore, the results will lead to modernization and an increase in the share of innovative organ-replacing technologies in the health care system.

## 2. Explanatory note

#### 1. General information

- 1.1. Name of the topic of the scientific, scientific and technical program "Development of innovative technologies for the treatment of pulmonary and heart failure to prolong human's life"
  - 1.3. Location of the program. ~The Republic of Kazakhstan, Nur-Sultan.
- 1.4. Estimated start and end date of the program, its duration in months. 2021 2023 years, 36 months.
- 1.5. Organization applying for the program. Non-profit JSC "National Research Center for Cardiac Surgery".
- 1.6. Executors of the program. Non-profit JSC «National Research Center for Cardiac Surgery».
- 1.7. The requested amount of targeted program financing for the entire duration of the program is 240 265 thousand tenge, 2021 84 107 thousand tenge, 2022 84 817 thousand tenge, 2023 71 340 thousand tenge.
- 1.8. Key words characterizing the sector and the direction of the program for the selection of independent experts. Anesthesiology. Cardiothoracic surgery. Nephrology. Perfusion. Efferentology.

#### 2. The general concept of the program.

## 2.1. Introductory part.

Non-profit JSC «National Research Center for Cardiac Surgery» (hereinafter – Non-profit JSC "NRCCS") is a research center that implements a program for the treatment of patients with chronic heart failure (CHF) and pulmonary failure (PF) in the terminal stage, including orthotopic transplantation of the heart and lungs, mechanical support of blood circulation

Scientific supervisor of the program - Yuriy Vladimirovich Pya - Director for Surgery and Science of the Non-profit JSC «NRCCS», Associate Professor, Doctor of Medical Sciences, cardiac surgeon of the highest category.

Scientific co-director of the program - Timur Dostaevich Lesbekov - Non-profit JSC «National Research Center for Cardiac Surgery», candidate of medical sciences, cardiac surgeon of the highest category.

The implementation of this program will improve organ recovery, reduce postoperative complications, reduce postoperative mortality and improve the quality of life of patients with pulmonary and heart failure.

## 2.2. The purpose of the program.

Development of new treatments heart and pulmonary failure using organ-replacing technologies.

Development of a clinical protocol and implementation of treatment methods into clinical practice heart and pulmonary failure using organ-replacing technologies.

# 2.3. Objectives of the program.

# Task 1. Assessment the results of the use of extracorporeal life support systems in the treatment of pulmonary and / or heart failure.

- Subtask 1.1. Assessment of the restoration of organ function during extracorporeal life support systems using extracorporeal hemocorrection.
- Subtask 1.2. Assessment of the normalization of the body's immune response and restoration of organ function during extracorporeal life support systems using an extracorporeal cytokine adsorber.

# Task 2. Studying the restoration of organ function during implantation of the left ventricular assist device as an organ-replacing aid in heart failure.

- Subtask 2.1. Assessment of the restoration of organ function during implantation of the left ventricular assist device with the use of extracorporeal hemocorrection.
- Subtask 2.2. Assessment of the normalization of the body's immune response and restoration of organ function upon implantation of the left ventricular assist device using an extracorporeal cytokine adsorber.

# Task 3. Studying the restoration of organ function during the implantation of the total artificial heart as an organ-replacing aid in case of heart failure.

- Task 3.1. Assessment of normalization of organ function restoration during implantation of the total artificial heart with the use of extracorporeal hemocorrection.
- Task 4. Studying the restoration of organ function during operations in conditions of the long-term cardiopulmonary bypass.

Task 4.1. Assessment of the restoration of organ function during operations with long-term cardiopulmonary bypass, hypothermia and circulatory arrest, with the use of extracorporeal hemocorrection.

Task 4.2. Assessment of the restoration of organ function during operations with long-term cardiopulmonary bypass, hypothermia and circulatory arrest using an extracorporeal cytokine adsorber.

# Task 5. Improvement of the method of implantation of organ-replacing technologies to reduce complications in the treatment of heart and pulmonary failure.

# 3. Scientific innovativeness and significance of the program.

Organ replacement technologies are increasingly being used in the treatment of endstage pulmonary and heart failure to prolong human life. Severe refractory cardiogenic shock, refractory ventricular arrhythmia, active cardiopulmonary resuscitation in cardiac arrest and acute or decompensated right heart failure, sepsis, pulmonary and multiple organ failure.

Careful patient selection and consideration of possible complications are key factors in optimizing the treatment of patients in this category. Well-defined pathways for medical care to centers capable of delivering heart and lung support replacement therapy (e.g., durable ventricular assist device or heart transplant) is essential to provide high-level patient care, stabilized with extracorporeal life support, and the ability to wean from the device. Ultimately, the concentration of the most complex care in large centers of our country with developed cardiac surgery and anesthetic capabilities can be a way to significantly improve the care of this group of patients.

Despite advances in mechanical ventilation, severe acute pulmonary distress syndrome (APDS) is associated with high morbidity and mortality rates ranging from 26% to 58%. Extracorporeal life sustaining system is a procedure for long-term cardiopulmonary bypass and oxygen saturation of the blood outside the body, used in patients with acutely developed and potentially reversible pulmonary and / or heart failure, whose treatment does not respond to maximum standard therapy. The Heart-Lung Sustaining System is a complex network that provides oxygenation and ventilation and allows the lungs to rest and recover from pulmonary failure while minimizing the iatrogenic lung damage caused by the ventilator. In intensive care in the conditions of an extracorporeal life support system. In 2011, the National Research Center for Cardiac Surgery Non-profit JSC launched a program to provide extracorporeal life support system in Kazakhstan, and in 2016 Non-profit JSC «NRCCS» has entered to the global ELSO register (Extracorporeal Life Support Organization).

The constant increase in the number of patients with CHF is associated with both an increase in the life expectancy of patients and a decrease in mortality among patients with a complicated course of acute myocardial infarction, heart defects, etc. The most common causes leading to the development of CHF are arterial hypertension, coronary heart disease and myocardial infarction. The gold standard for treatment of patients with end-stage heart failure, tolerant to drug therapy is heart transplantation.

Deficiency of donor organs remains the most important factor holding back the development of lung and heart transplantation all over the world and in our country. Left ventricular assist device (LVAD) implantation is a bridge to heart transplantation, which improves the quality and duration of life by improving blood circulation in most patients with chronic heart failure [1]. In recent studies, it was shown that the 1-year survival rate of patients after implantation of mechanical blood circulation support devices as a "bridge to transplantation" (BTT - bridge to transplantation) was 85%, and the 2-year survival rate in patients with ventricular assist device as " final treatment "(" DT - destination therapy ") - 76% [2]. It was also noted that patients with LVAD support improve functional status and quality of life [2].

A Total Artificial Heart is a form of mechanical circulatory support in which the patient's ventricles and valves are removed and replaced with an artificial heart. Currently, a fully artificial heart is implanted in the terminal stage of biventricular heart failure as a "bridge" to heart transplantation. However, given the increasing global burden of cardiovascular disease and congenital heart disease with heart failure, the number of end-stage heart failure patients awaiting heart transplants now far outnumbers the available hearts. As a result, the use of mechanical circulatory support, including a fully artificial heart, is growing exponentially.

Sepsis, septic shock, and systemic inflammatory response syndrome are life-threatening conditions resulting from a systemic response. Dysregulation can lead to multiple organ dysfunctions [30-36].

While sepsis and septic shock are infectious in origin, systemic inflammatory response syndrome (SIRS) can also have noninfectious triggers such as open heart bypass surgery, ex vivo heart / lung perfusion, extracorporeal life support, and mechanical circulatory support. It should be noted that mortality in SIRS, septic shock and sepsis reaches 7, 16, and 40%, accordingly [37-45]. According to Sepsis-3 2016, the new definition has two categories: sepsis and septic shock [46-49]. Previous definitions of sepsis, published in 1992, have

highlighted the role of systemic inflammatory response syndrome (SIRS) as a key element in the definition of sepsis.

In order to improve the results of implantation of mechanical devices, patients on the extracorporeal life support system and septic patients before surgery, various techniques are used to reduce the syndrome of systemic inflammatory response, immunocorrection, and others. To date, there are many ways to prevent the development of a systemic inflammatory response by removing leukocytes from the bloodstream by including a filter with a special screen in the perfusion circuit to remove leukocytes and prevent the latter from entering the systemic circulation [9].

The most effective is the method of extracorporeal hemadsorption, intended for additional therapy of patients with an increased level of cytokines in conditions of the systemic inflammatory response syndrome, in which a patient with acute pulmonary distress syndrome and cardiogenic septic shock against the background of an extracorporeal system has additional life support in the circuit of the apparatus for the veno-venous hemofiltration, an extracorporeal cytokine adsorber system was installed, designed to eliminate a wide range of inflammatory mediators, as well as various proteins and metabolites [55-61].

There are some new data showing that the use of an extracorporeal cytokine adsorber for long periods of cardiopulmonary bypass surgery (> 120 minutes) may be useful for preventing SIRS and reducing cytokine levels in patients have overcome by elective heart surgery [62-68].

In this study, methods will be developed to restore the function of affected organs before and / or after mechanical support of blood circulation (implantation of a completely artificial heart, implantation of an artificial left ventricle, an extracorporeal life support system) in combination with the use of an extracorporeal cytokine adsorber, which will improve the results of surgical treatment of patients with terminal heart and pulmonary failure.

New methods developed for restoring the function of affected organs after implantation of an artificial left ventricle, a completely artificial heart, an extracorporeal life support system will be of high importance, both for Kazakhstan and for states with similar problems of donor organ deficiency, will also improve the effectiveness of surgical treatment and reduce the level of complications and mortality of patients on the extracorporeal life support system and septic patients.

The clinical study data will form the basis of practical protocols for the implantation of an artificial left ventricle, a fully artificial heart, an extracorporeal life support system, following which will improve organ recovery, reduce postoperative complications, improve the quality of life and reduce mortality after surgery.

#### 4. Research methods and ethical issues.

All patients admitted to Non-profit JSC "NRCCS" who meet the study criteria (patients on an extracorporeal life support system, mechanical circulatory support, surgery on the aortic arch) will be included in the study after obtaining a signed informed consent. Participants will be randomized into 2 groups in a 1: 1 division.

**Intervention team # 1** using an extracorporeal hemoperfusion device Jafron (Zhuhai Jafron Biomedical, China) (50 patients) in subgroups: A (n = 10) - patients on extracorporeal life support systems with heart failure; B (n = 10) - patients on extracorporeal life support systems with pulmonary failure; C (n = 5) - patients with implantation of a left ventricular accessory device; D (n = 25) - during operations with prolonged artificial circulation, hypothermia and circulatory arrest.

**Intervention team # 2** using extracorporeal cytokine, CytoSorb (CytoSorbents Corporation, Monmouth Junction, NJ, USA) (50 patients) in subgroups: A (n = 10) - patients on extracorporeal life support systems in heart failure; B (n = 10) - patients on extracorporeal life support systems with pulmonary failure; C (n = 5) - patients with implantation of a left ventricular accessory device; D (n = 25) - during operations with prolonged artificial circulation, hypothermia and circulatory arrest.

# Retrospective analysis of patients who received a fully artificial heart.

The duration of the intervention in each group will be 72 hours. Each Jafron / CytoSorb Removal Column can be used within 24 hours, so all patients in 2 groups use 3 filters during the study.

Researchers will collect demographic, clinical and laboratory data from patients before, during and after surgery.

The incidence of early cellular or humoral rejection, the duration of ventilation, intensive care and hospital stay, the use of vasopressors and inotropes in the perioperative period, and the incidence of perioperative complications and survivals will be documented.

The level of cytokines (IL-1, IL-6, IL-8, IL-10, tumor necrosis factor alpha) and complements will be determined before, during and after the use of the extracorporeal life support system for heart and pulmonary failure; surgery on the aortic arch, patients on mechanical circulatory support, if investigators find a corresponding difference between the two groups in terms of clinical variables.

# Study design.

Study type: interventional (clinical study)

Set of participants: 100 participants

Distribution: randomized

Interventional model: parallel

Masking: no

Primary Goal: Treatment

| Intervention team (1 group) | Intervention / treatment (device) |
|---|---|
| Extracorporeal hemoperfusion device will be | HA330 - Jafron Biomedical Co., Ltd., China |
| installed in the device of the extracorporeal | - extracorporeal hemocorrection, which is |
| life support system for heart failure | based on the removal of cytokines from |
| (10 patients) | whole blood by sorption on a special |
| | hemoadsorbent due to the peculiarities of its |
| | porous structure and inner surface, which is |
| | indicated in conditions where cytokine levels |
| | are extremely elevated. |
| Extracorporeal hemoperfusion device will be | HA330 - Jafron Biomedical Co., Ltd., China |
| installed in the device of the extracorporeal | - extracorporeal hemocorrection, which is |
| life support system for pulmonary failure | based on the removal of cytokines from |
| (10 patients). | whole blood by sorption on a special |
| | hemabsorbent due to the peculiarities of its |
| | porous structure and inner surface, which is |
| | indicated in conditions where cytokine levels |
| | are extremely elevated. |
| An extracorporeal hemoperfusion device will | HA330 - Jafron Biomedical Co., Ltd., China |
| be installed in patients before / during the | - extracorporeal hemocorrection, which is |
| implantation of a left ventricular assist device | based on the removal of cytokines from |
| (5 patients). | whole blood by sorption on a special |
| | hemoadsorbent due to the peculiarities of its |
| | porous structure and inner surface, which is |
| | indicated in conditions where cytokine levels |
| | are extremely elevated. |
| An extracorporeal hemoperfusion device will | HA330 - Jafron Biomedical Co., Ltd., China |

be installed in patients during operations with - extracorporeal hemocorrection, which is prolonged cardiopulmonary based on the removal of cytokines from bypass, hypothermia and circulatory arrest. (25 whole blood by sorption on a special hemoadsorbent due to the peculiarities of its patients). porous structure and inner surface, which is indicated in conditions where cytokine levels are extremely elevated. **Intervention team (2 groups)** CytoSorb (CytoSorbents Corp., USA) - an Extracorporeal hemoperfusion device will be installed in the device of the extracorporeal extracorporeal cytokine adsorber life support system for heart failure. biocompatible polymer with high adsorption (10 patients) capacity, which is indicated in conditions where cytokine levels are extremely elevated. Extracorporeal hemoperfusion device will be CytoSorb (CytoSorbents Corp., USA) - an installed in the device of the extracorporeal extracorporeal cytokine adsorber is life support system for pulmonary failure. biocompatible polymer with high adsorption (10 patients) capacity, which is indicated in conditions where cytokine levels are extremely elevated. An extracorporeal hemoperfusion device will CytoSorb (CytoSorbents Corp., USA) - an be installed in patients before / during the extracorporeal cytokine adsorber implantation of a left ventricular assist device biocompatible polymer with high adsorption (5 patients) capacity, which is indicated in conditions where cytokine levels are extremely elevated. An extracorporeal hemoperfusion device will CytoSorb (CytoSorbents Corp., USA) - an be installed in patients during operations with extracorporeal cytokine adsorber is a prolonged cardiopulmonary bypass, biocompatible polymer with high adsorption hypothermia and circulatory arrest. (25 capacity, which is indicated in conditions where cytokine levels are extremely elevated. patients)

#### **Performance evaluation criterias**

| | Extracorporeal life support system with pulmonary and / or heart failure |
|---|---|
| Prima | ry results |

| 1 | Cytokine response [Time: 24-48 hours] |
|---|---|
| | The level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-8, IL-10, tumor |
| | alpha-factor) before the implantation, 2 hours after the start of ECMO support, |
| | explantation of ECMO, 24 hours after explantation of ECMO. |
| 2 | SOFA-Score [Time Frame: 24, 48, 72 hours] |
| | Sequential Organ Failure Assessment Score at 24, 48, 72 h (values from 6 to 24, |
| | where the higher values explain higher disease severity) |
| 3 | Difference of mean arterial pressure [Time Frame: 24, 48, 72 hours] |
| | Comparison of mean arterial pressure at 24, 48, 72 hours between between two |
| | interventions (CytoSorb and Jafron) |
| 4 | Difference of CVP [Time Frame: 24, 48, 72 hours] |
| | Comparison of CVP at 24, 48, 72 hours between between two interventions |
| | (CytoSorb and Jafron) |
| 5 | Serum lactate [ Time Frame: 24, 48, 72 hours ] |
| | Level of serum lactate at 24, 48, 72 h |
| 6 | Days on ventilator, vasopressor and renal replacement therapy [ Time Frame: until |
| | day 30 post-surgery ] |
| | Total days on ventilator, vasopressor and renal replacement therapy within 30 days |
| | post-surgery will be assessed |
| 7 | Doses of vasopressors and / or inotropes (µg / h / kg bodyweight) [Time: first 72 |
| | hours] |
| Secon | dary results |
| 1 | Inflammatory response - The level of C-reactive protein (CRP) [Time: 24-48 hours] |
| | The level of C-reactive protein (CRP) before the start of ECMO, 2 hours after the |
| | implantation of ECMO, during ECMO, 24 hours after ECMO explantation. |
| 2 | Inflammatory response - The level of leukocytes [Time: 24-48 hours] |
| | The level of leukocytes before the start of ECMO, 2 hours after the implantation of |
| | ECMO, during ECMO, 24 hours after ECMO explantation. |
| 3 | Inflammatory response - The level of procalcitonin [Time: 24-48 hours] |
| | The level of procalcitonin before the start of ECMO, 2 hours after the implantation of |
| | ECMO, during ECMO, 24 hours after ECMO explantation. |
| 4 | Level of leukocyte [Time: 24-48 hours] |
| | Level of leukocyte cells in the bloodstream at 24, 48 hours. |

| 5 | Application and dosage of vasopressors [Deadline: first 48 hours] |
|---|---|
| | Incidence of application and level of dosage of vasopressors on days 2 and 3 after |
| | surgery; |
| 6 | Application and dosage of inotropes [Deadline: first 48 hours] |
| | Incidence of application and level of dosage of inotropes on days 2 and 3 after |
| | surgery; |
| Long- | term results |
| 1 | Length of stay in the intensive care unit [Duration: first 48 hours] |
| 2 | Length of hospital stay [Term: up to 1 month]; |
| 3 | 30 day survival rate. |

| | Patients with left ventricular assist device implantation |
|---|---|
| Primo | ary results |
| 1 | Difference of Cytokine response [Time: 24-48 hours] |
| | Level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-8, IL-10, tumor |
| | necrosis factor-alfa, procalcitonin) |
| 2 | Doses of vasopressors and / or inotropes (µg / h / kg bodyweight) |
| | [Deadline: first 72 hours] |
| 3 | Renal function [Time: first 72 hours] creatinine level |
| 4 | Lactate level [Time: first 72 hours] |
| Secon | idary results |
| 1 | Inflammatory response - The level of C-reactive protein (CRP) [Time: 24-48 hours] |
| | The level of C-reactive protein (CRP) before the start of the operation, 2 hours after |
| | the start of the operation, when the operation is turned off, 24 hours after the |
| | shutdown of the operation |
| 2 | Inflammatory response - The level of leukocytes [Time: 24-48 hours] |
| | The level of leukocytes before the start of the operation, 2 hours after the start of |
| | the operation, when the operation is turned off, 24 hours after the shutdown of the |
| | operation |
| 3 | Inflammatory response - The level of procalcitonin [Time: 24-48 hours] |
| | The level of procalcitonin before the start of the operation, 2 hours after the start of |
| | the operation, when the operation is turned off, 24 hours after the shutdown of the |
| | operation |

| 4 | Application and dosage of vasopressors [Deadline: first 48 hours] |
|---|---|
| | Incidence of application and level of dosage of vasopressors on days 2 and 3 after |
| | surgery; |
| 5 | Application and dosage of inotropes [Deadline: first 48 hours] |
| | Incidence of application and level of dosage of inotropes on days 2 and 3 after |
| | surgery; |
| Long- | term results |
| 1 | Length of stay in the intensive care unit [Duration: first 48 hours] |
| 2 | Length of hospital stay [Term: up to 1 month]; |
| 3 | 30 day survival rate. |

| | For operations with prolonged cardio pulmonary bypass, hypothermia and |
|---|---|
| | circulatory arrest |
| Primo | ary results |
| 1 | Cytokine response [Time: 24-48 hours] |
| | Difference of Cytokine response [Time: 24-48 hours] |
| | Level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-8, IL-10, tumor |
| | necrosis factor-alfa, procalcitonin, C-reactive protein) |
| 2 | SOFA-Score [Time Frame: 24, 48, 72 hours] |
| | Sequential Organ Failure Assessment Score at 24, 48, 72 h (values from 6 to 24, |
| | where the higher values explain higher disease severity) |
| 3 | Difference of mean arterial pressure [Time Frame: 24, 48, 72 hours] |
| | Comparison of mean arterial pressure at 24, 48, 72 hours between between two |
| | interventions (CytoSorb and Jafron) |
| 4 | Difference of CVP [Time Frame: 24, 48, 72 hours] |
| | Comparison of mean arterial pressure at 24, 48, 72 hours between between two |
| | interventions (CytoSorb and Jafron) |
| 5 | Level of Serum lactate [ Time Frame: 24, 48, 72 hours ] |
| | Comparison of mean arterial pressure at 24, 48, 72 hours between between two |
| | interventions (CytoSorb and Jafron) |
| Secor | ndary results |
| 1 | Inflammatory response - The level of C-reactive protein (CRP) [Time: 24-48 hours] |
| | The level of C-reactive protein (CRP) before the cardiopulmonary bypass 2 hours |

| | after the cardiopulmonary bypass, when the cardiopulmonary bypass is turned off, |
|---|---|
| | 24 hours after the cardiopulmonary bypass. |
| 2 | Inflammatory response - The level of leukocytes [Time: 24-48 hours] |
| | The level of leukocytes before the cardiopulmonary bypass 2 hours after the |
| | cardiopulmonary bypass, when the cardiopulmonary bypass is turned off, 24 hours |
| | after the cardiopulmonary bypass. |
| 3 | Inflammatory response - The level of procalcitonin [Time: 24-48 hours] |
| | The level of procalcitonin before the cardiopulmonary bypass 2 hours after the |
| | cardiopulmonary bypass, when the cardiopulmonary bypass is turned off, 24 hours |
| | after the cardiopulmonary bypass. |
| 4 | Application and dosage of vasopressors [Deadline: first 48 hours] |
| | Incidence of application and level of dosage of vasopressors on days 2 and 3 after |
| | surgery; |
| 5 | Application and dosage of inotropes [Deadline: first 48 hours] |
| | Incidence of application and level of dosage of inotropes on days 2 and 3 after |
| | surgery; |
| Long- | ong-term results |
| 1 | Length of stay in the intensive care unit [Duration: first 48 hours] |
| 2 | Length of hospital stay [Term: up to 1 month]; |
| 3 | 30 day survival rate. |

## Statistical research

- 1) statistical data processing
- 2) comparison and analysis of initial data

After data acquisition, statistical analysis will be performed using SPSS Statistics version 22. For quantitative data, the nonparametric Mann-Whitney Yu test and parametric test will be performed, and for qualitative studies, the nonparametric Fisher's exact test and the parametric  $\chi^2$  test will be performed. Also, logistic regression for categorical outcomes and survival analyzes (non-parametric Kaplan-Meyer and parametric Cox regression) will be performed.

Age: 18 years and older

Gender: All

**Inclusion of healthy volunteers:** Not

| Groups | Inclusion criteria | Exclusion criteria |
|---|---|---|
| Patients on an | • Implantation of intravenous | Age less than 18 years old |
| extracorporeal life | ECMO | • Terminal hepatic or renal |
| support system with | • Hemodynamic support with | failure just before the |
| heart failure | vasopressors and / or tonics; | procedure |
| | • Procalcitonin level ≥ 1 ng / ml; | • Patient's written refusal to |
| | • Invasive hemodynamic | participate in the study |
| | monitoring; | |
| | Written informed consent. | |
| Patients on an | IV ECMO implantation | Age less than 18 years old |
| extracorporeal life | • High levels of venous and | • Terminal hepatic or renal |
| support system with | arterial CO2 (CO2> 50 | failure just before the |
| pulmonary failure | mmHg), | procedure |
| | | • Patient's written refusal to |
| | • Low paO2, SvO2, SpO2. | participate in the study |
| | • Invasive hemodynamic | |
| | monitoring; | |
| | Written informed consent. | |
| Patients with left | LVAD implantation | Age less than 18 years old |
| ventricular assistive | Biventricular heart failure IV | Acute hepatic or renal failure |
| device implantation | • INTERMACS I-III | just before the procedure |
| | • Hemodynamic support with | • Patient's written refusal to |
| | vasopressors and / or tonics; | participate in the study |
| | • Procalcitonin level ≥ 0.1 ng / ml; | |
| | • Invasive hemodynamic | |
| | monitoring; | |
| | Written informed consent. | |
| Patients in operations | Hemodynamic support with | Age less than 18 years old |
| with prolonged artificial | vasopressors and / or tonics; | • Terminal hepatic or renal |
| circulation, hypothermia | • Bypass duration> 120 minutes | failure just before the |
| and circulatory arrest | • Hypothermia ≤ 25 0C | procedure |
| | Circulatory arrest | • Patient's written refusal to |

| • Procalcitonin level ≥ 1 ng / ml; | | participate in the study |
|------------------------------------|-------------|--------------------------|
| • Invasive | hemodynamic | |
| monitoring; | | |
| • Written informed of | consent. | |

The study will be conducted in accordance with the international standards Good Clinical Practice, Joint Commission International, scientific ethics (Declaration of Helsinki), as well as the Order of the Minister of Health of the Republic of Kazakhstan dated December 11, 2020 No. 248 "On approval of the rules for conducting clinical trials of drugs and medical devices, clinical laboratory testing of medical devices for diagnostics outside of a living organism (in vitro) and requirements for clinical bases and provision of public services. Issuance of a permit for conducting a clinical trial and (or) testing of pharmacological and medicinal products, medical devices. "The study will also take place in accordance with the recommendations of the Local Ethics Commission at Non-profit JSC «NRCCS». All patients will receive a voluntary informed consent of the established form with permission to use clinical data for scientific purposes. In addition, the research will be strictly monitored by the researchers to ensure that it is free from plagiarism, falsification and fabrication of data in order to achieve the highest ethical conduct of the research. The resulting patient data will be strictly confidential with ensuring privacy through strictly limited access to data, de-identification of data and destruction after the end of the study.

# 5. Research team and program management

| No | Full name | Main place of | | Employment | Project work period (months) | | |
|---|---|---|---|---|---|---|---|
| | (degree, academic title) | work, position | Role in the program | | 1st year | 2nd year | 3rd year |
| | | | Leader | | | | |
| | | | Scientific supervisor of the project. | | | | |
| | | Non-profit JSC | General project management, | | | | |
| 1 | Pya | "NRCCS" | definition of the vision and | Part-time | 12 | 12 | 12 |
| 1 | Yuri | Director of Science | direction of the project, | ran-ume | | | |
| | Vladimirovich | and Surgery | participation in the analysis of | | | | |
| | | | results, participation in the | | | | |
| | | | preparation of publications | | | | |
| | | Non-profit JSC | Co-leader | | | | |
| | | "NRCCS" | General project management, | | | | |
| | Lesbekov | Head of the | definition of the vision and | | | | |
| 2 | Timur | Department of | direction of the project, | Part-time | 12 | 12 | 12 |
| | Dostaevich | Cardiac Surgery | participation in the analysis of | | | | |
| | | | results, participation in the | | | | |
| | | | preparation of publications | | | | |
| 3 | Kaliev | Non-profit JSC | Leading researcher | Part-time | | | |

| | Rymbay | "NRCCS" | Selection of patients, analysis of | | | | |
|---|---|---|---|---|---|---|---|
| | Bolatovich | Head of the | clinical data, development of a | | | | |
| | | operating | quality of life questionnaire. | | 12 | 12 | 12 |
| | | department with a | Participation in the analysis of | | | | |
| | | laboratory for | results and preparation of | | | | |
| | | circulatory support | publications, methods, including | | | | |
| | | | methods of prevention. | | | | |
| | | Non-profit JSC | Secondary researcher | | | | |
| | | "NRCCS" | Selection of patients, analysis of | | | | |
| | Nurmykhametova<br>Zhuldyz<br>Askarovna | Physician | clinical data, development of a | | | | |
| 4 | | perfusionist of the | quality of life questionnaire. | Part-time | 12 | 12 | 12 |
| 4 | | operating | Participation in the analysis of | | | | |
| | | department with a | results and preparation of | | | | |
| | | laboratory for | publications, methods, including | | | | |
| | | circulatory support | methods of prevention | | | | |
| | | | Secondary researcher | | | | |
| | | Non-profit JSC | Selection of patients, analysis of | | | | |
| 5 | Kuanyshbek | "NRCCS" | clinical data, development of a | Part-time | | | |
| 3 | Aydin Sayatovich | Head of the | quality of life questionnaire. | Part-time | 12 | 12 | 12 |
| | | Department of | Participation in the analysis of | | | | |
| | | Anesthesiology, | results and preparation of | | | | |

| | | Reanimation and Intensive Care | publications, methods, including methods of prevention | | | | |
|---|---|---|---|---|---|---|---|
| 6 | Dzhabaeva<br>Nilufar<br>Amirbekovna | Non-profit JSC "NRCCS" Doctor nephrologist Extracorporeal hemocorrection laboratories | SNS Selection of patients, analysis of clinical data, development of a quality of life questionnaire. Participation in the analysis of results and preparation of publications, methods, including methods of prevention | Part-time | 12 | 12 | 12 |
| 7 | Faizov<br>Linar<br>Renatovich | Non-profit JSC "NRCCS" Physician perfusionist of the operating department with a laboratory for circulatory support | SNS Selection of patients, analysis of clinical data, development of a quality of life questionnaire. Participation in the analysis of results and preparation of publications, methods, including methods of prevention | Part-time | 12 | 12 | 12 |
| 8 | Position | | Economic calculations, preparation of interim and annual reports | Part-time | | | |

| | | | | | 12 | 12 | |
|---|---|---|---|---|---|---|---|
| | | | | | | | 12 |
| 9 | Iskakova<br>Ainel<br>Talgatovna | Non-profit JSC "NRCCS" Chief Specialist Department of Science | Organizational project management, preparation of semi-annual acts, reports. | Part-time | 12 | 12 | 12 |
| 10 | Position | | Statistical processing of the obtained research data | Part-time | | | |
| 11 | Position | | Statistical processing of the obtained research data | Part-time | | | |

In total, 11 specialists in the field of cardiac surgery, perfusion, cardiology, anesthesiology, efferentology, and public health are involved in the project.

Principal Investigator - Yuriy Vladimirovich Pya - Director for Surgery and Science of the National Research Center for Cardiac Surgery, a graduate of the 2nd Moscow State Medical Institute named after V.I. NI Pirogova, international cardiac surgeon, associate professor, doctor of medical sciences. Winner of a number of state awards, including the Order of the Republic of Kazakhstan "Parasat", "Doctor of the Year 2012", the honorary title "Kazakhstan Enbek Eri". The supervisor will be involved throughout the entire research period. According to Scopus, the Hirsch index - 10, Author ID in Scopus - 7801690331. Proncipal Investigator of the projects:

- 1. Scientific project Committee of Science of the Ministry of education and science of Republic of Kazakhstan 2018-2020 on the topic "Study of the effectiveness of a new method of conditioning for the preservation of the donor heart";
- 2. Scientific program Targeted program financing of the Ministry of Health of the Republic of Kazakhstan 2017-2019 on the topic "New molecular genetic methods of pre-symptomatic diagnostics and methods of treatment of a number of significant diseases", Surgical treatment of CHF;
- 3. Y. Pya, A. Medressova, S. Bekboыsynov, dated August 25, 2020, No. US 10,751,456 B2, METHOD OF IMPLANTATION OF LEFT VENTRICULAR MECHANICAL ASSIST DEVICE HEARTMATE III (US Patent Office);
- 4. Y. Pya, A. Medressova, S. Bekbossynov, dated November 16, 2020, No. 201800238 Method of implantation of a device for mechanical support of the left ventricle HEARTMATE 3 (Eurasian Patent Office).

Co-head of the program - Timur Dostaevich Lesbekov, Candidate of Medical Sciences, Head of the Department of Cardiac Surgery, Non-profit JSC «NRCCS». According to Scopus, the Hirsch index - 2, the Author ID in Scopus - 6505523476.

Kaliev Rymbay Bolatovich - head of the operating department with the laboratory of auxiliary blood circulation, Non-profit JSC «NRCCS». According to Scopus, Hirsch index is 3, Author ID in Scopus - 57053326800.

Kuanyshbek Aydin Sayatovich - Head of the Department of Anesthesiology, Reanimation and Intensive Care of the Non-profit JSC «NRCCS». According to Scopus, Hirsch index - 1, Author ID in Scopus -57221294150.

Nurmykhametova Zhuldyz Askarovna - doctor perfusionist of the operating department with a laboratory for auxiliary circulation of the Non-profit JSC «NRCCS». According to Scopus, Hirsch index - 1, Author ID in Scopus -57221292855.

Faizov Linar Renatovich - doctor perfusionist of the operating department with the laboratory of auxiliary circulation of the Non-profit JSC «NRCCS». According to Scopus, Hirsch index - 2, Author ID in Scopus - 57194181173.

# List of international publications (last):

| 1 | Medressova, A., Faizov, L., Kuanyshbek, A., Kaliyev, R., Myrzakhmetova, G., la |
|---|---|
| | Fleur, P., Pya, Y. Successful heart transplantation after 17 h ex vivo time using the |
| | Organ Care System—3 years follow-up//Journal of Cardiac Surgery, 2021 (in |
| | press) (52 percentile, Scopus) |
| 2 | Zimpfer, D., Gustafsson, F., Potapov, E., Pya, Y., Schmitto, J., Berchtold-Herz, |
| | M., Garbade, J. (2020). Two-year outcome after implantation of a full |
| | magnetically levitated left ventricular assist device: Results from the ELEVATE |
| | registry. European Heart Journal, 41(39), 3801-3809. |
| | doi:10.1093/eurheartj/ehaa639 (99 percentile, Scopus) |
| 3 | Pya, Y., Netuka, I., Latremouille, C., Bekbossynova, M., Medressova, A., |
| | Bekbossynov, S., Salov, R., & Hetzer, R. (2020). CARMAT total artificial heart |
| | implantation: report on the first successful clinical experience as bridge to heart |
| | transplantation. Cardiovascular Diagnosis And Therapy, 0. doi:10.21037/cdt-20- |
| | 353 (63 percentile, Scopus) |
| 4 | Mirza, Kiran & Gustafsson, F. & Pya, Y. & Shaw, S. & Diegeler, A. & Netuka, I. |
| | & Lavee, Jacob & Garbade, Jens & Morshuis, M. & Heatley, J. & Saeed, Diyar & |
| | Potapov, Evgenij & Schmitto, Jan & Zimpfer, Daniel. (2019). Atrial Fibrillation is |
| | a Predictor of Poor Physical Capacity 6 Months after Implantation of a Full |
| | Magnetically Levitated Left Ventricular Assist Device: An Analysis from |
| | ELEVATE. The Journal of Heart and Lung Transplantation. 38. S45. |
| | 10.1016/j.healun.2019.01.095. (99 percentile, Scopus) |
| 5 | Netuka, I. & Pya, Y. & Zimpfer, Daniel & Potapov, E. & Garbade, Jens & Rao, V. |
| | & Morshuis, M. & Marasco, S. & Beyersdorf, F. & Gazzola, C. & Sood, P. & |
| | Schmitto, Jan. (2020). First Long-Term 5-years experience with the HeartMate 3 |
| | LVAS in Multicentric Clinical Trial. The Journal of Heart and Lung |

| | Transplantation. 39. S184. 10.1016/j.healun.2020.01.768. (99 percentile, Scopus) |
|---|---|
| 6 | Loforte, Antonio & Gliozzi, G. & Potapov, E. & Mariani, Carlo & Schoenrath, |
| | Felix & Netuka, I. & Pya, Y. & Gummert, Jan & Meyns, B. & Pacini, Doreen & |
| | By, T.M.M.H. (2020). Concomitant Cardiac Procedures during Implantation of |
| | Long-Term Continuous-Flow LVADs: A European Registry for Patients with |
| | Mechanical Circulatory Support (EUROMACS) Analysis. The Journal of Heart |
| | and Lung Transplantation. 39. S122-S123. 10.1016/j.healun.2020.01.1009. (99 |
| | percentile, Scopus) |
| 7 | Kaliyev, R., Lesbekov, T., Bekbossynov, S. Samalavicius, R., Pya, Y. |
| | Comparison of Custodiol vs warm blood cardioplegia and conditioning of donor |
| | hearts during transportation with the organ care system//Journal of Cardiac |
| | Surgery, 2019, 34(10), с. 969-975 (52 процентиль, Scopus) |
| 8 | R. Kaliyev, S. Bekbossynov, Zh. Nurmykhametova. Sixteen-Hour Ex Vivo Donor |
| | Heart Perfusion During Long-Distance Transportation for Heart |
| | Transplantation//Artificial organs - 43(3), 2019, c. 319-320 (60 percentile, |
| | Scopus) |
| 9 | <u>Пя Ю.В., Калиев Р.Б., Лесбеков Т.Д.,</u> Бекбосынов С.Т., Капышев Т.С., |
| | Нурмыхаметова Ж.А., Смагулов Н.К., Аширов Ж.З., Фаизов Л.Р. Программа |
| | экстракорпоральной мембранной оксигенаций в Казахстане: ближайшие |
| | результаты // «Журнал им. акад. Б.В. Петровского Клиническая и |
| | экспериментальная хирургия» - №1-2017 г. С. 41-45 (6 percentile, Scopus) |
| 10 | <u>Пя Ю.В., Калиев Р.Б.,</u> Бекбосынов С.Т., <u>Лесбеков Т.Д., Нурмыхаметова Ж.А.,</u> |
| | Смагулов Н.К., Новикова С.П., Аширов Ж.З., Фаизов Л.Р., Медресова А.Т., |
| | Мурзагалиева М.О. Новый метод сохранения донорского сердца с |
| | использованием кровяной кардиоплегии и кондиционирования // «Журнал |
| | им. акад. Б.В. Петровского Клиническая и экспериментальная хирургия» - |
| | №3-2017 г. С. 54-60 (6 percentile, Scopus) |
| | <u>Пя Ю.В.</u> , Бекбосынов С.Т., Бекбосынова М.С., Куатбаев Е.М., <u>Лесбеков Т.Д.</u> , |
| | Калиев Р.Б., Джетыбаева С.К., Медресова А.Т., Нурмыхаметова Ж.А., |
| | Мурзагалиев М.У., Новикова С.П., Капышев Т.С.,Смагулов Н.К., Фаизов |
| | <u>Л.Р.</u> , <u>Вахрушев И.А.</u> , Андосова С.А., Мырзахметова Г.Ш., Надирбекова Г.Е., |
| | Шайсултанова С.Т., Дюсенбина Ж.С. Программа трансплантации сердца в |
| | эпоху механической поддержки кровообращения: опыт Республики |

| Казахстан | // | «Журнал | ИМ. | акад. | Б.В. | Петровского | Клиническая | И |
|---|---|---|---|---|---|---|---|---|
| эксперимен | нтал | ьная хирур | гия» - | №3-20 | 17 г. С | . 49-54(6 percei | ntile, Scopus) | |

# 8. Plan for the implementation of the program.

| P/ | Name of tasks and measures for their | Start of execution | Duration, | Expected results of the program implementation (in the context of tasks and activities), completion form | | |
|---|---|---|---|---|---|---|
| p<br>No. | No. implementation | (dd / mm / yy) | months | 1st year | 2nd year | 3rd year |
| 1 | 2 | 4 | 5 | 6 | 7 | 8 |
| 1 | Literature review on organ replacement technology in the treatment of patients with heart and pulmonary insufficiency | 2021 | 9 | A literature review on organ replacement technology in the treatment of patients with heart and lung failure will be obtained. | | |
| 1.1 | A review of the literature on the restoration of organ function when using extracorporeal life support systems as an organ-substituting aid for heart and pulmonary | 2021 | 3 | A review of the literature on the restoration of organ function using extracorporeal life support systems as an organ-substituting aid for heart and pulmonary failure will be obtained. | | |

| | failure. | | | |
|---|---|---|---|---|
| 1.2 | Literature review on implantation of mechanical circulatory devices using an extracorporeal cytokine adsorber | 2021 | 3 | A literature review on the implantation of mechanical circulatory devices using an extracorporeal cytokine adsorber will be obtained. |
| 1.3 | Literature review on the use of an extracorporeal cytokine adsorber in operations with prolonged artificial circulation, hypothermia and circulatory arrest | 2021 | 3 | A literature review will be obtained on the use of an extracorporeal cytokine adsorber in operations for reconstructing the aortic arch with hypothermia and cardiopulmonary bypass. |
| 2 | Based on the literature review, conduct a comparative assessment of the application of methods of extracorporeal hemoadsorption in | 2021 | 9 | Comparative evaluation will be carried out on the application of methods of extracorporeal hemoadsorption in pulmonary and heart failure |

| | pulmonary and heart | | | | | |
|---|---|---|---|---|---|---|
| | failure | | | | | |
| 3 | Patient recruitment | 2021 | | Patient recruitment for the study will begin | Patient recruitment will continue | Patient recruitment will continue |
| 3.1 | Recruiting of patients using extracorporeal life support systems as an organ-substituting aid for heart and pulmonary failure. | 2021 | 36 | Recruiting of patients using extracorporeal life support systems as an organ-substituting aid for heart and pulmonary failure. | Recruiting of patients when using extracorporeal life support systems, as an organ-substituting aid, with heart and pulmonary failure will continue | Recruiting of patients when using extracorporeal life support systems, as an organsubstituting aid, with heart and pulmonary failure will continue |
| 3.2 | Recruiting of patients for implantation of mechanical circulatory devices using an extracorporeal cytokine adsorber | 2021 | 36 | Recruiting will begin patients with implantation of mechanical circulatory devices using an extracorporeal cytokine adsorber | Recruiting patients for implantation of mechanical circulatory devices using an extracorporeal cytokine adsorber will continue | Recruiting patients for implantation of mechanical circulatory devices using an extracorporeal cytokine adsorber will continue |
| 3.3 | Recruiting of patients for hypothermia and cardiopulmonary bypass reconstruction with an extracorporeal cytokine | 2021 | 36 | Will be started recruiting of patients for reconstructions of the aortic arch with hypothermia and cardiopulmonary bypass | Recruiting of patients for hypothermia and cardiopulmonary bypass reconstruction with an extracorporeal cytokine | Recruiting of patients for hypothermia and cardiopulmonary bypass reconstruction with an extracorporeal cytokine |

| | adsorber | | | using an extracorporeal | adsorber will continue | adsorber will continue |
|---|---|---|---|---|---|---|
| | | | | cytokine adsorber | | |
| 4 | Collection of laboratory | 2021 | 36 | There will be a collection | There will be a collection | There will be a collection |
| - | and clinical data | 2021 | 30 | laboratory and clinical data | laboratory and clinical data | laboratory and clinical data |
| | Collection of laboratory | | | There will be a collection | There will be a collection | There will be a collection |
| | and clinical data, blood | | | laboratory and clinical data, | laboratory and clinical data, | laboratory and clinical data, |
| | sampling for pro- and | | | blood sampling for pro- and | blood sampling for pro- and | blood sampling for pro- and |
| | anti-inflammatory | | | anti-inflammatory cytokines, | anti-inflammatory cytokines, | anti-inflammatory cytokines, |
| | cytokines, assessment of | | | assessment of organ | assessment of organ | assessment of organ |
| 4.1 | organ dysfunction, dose | 2021 | 36 | dysfunction, dose of | dysfunction, dose of | dysfunction, dose of |
| 1.1 | of vasopressors after | 2021 | | vasopressors after | vasopressors after | vasopressors after |
| | implantation of | | | implantation of | implantation of | implantation of extracorporeal |
| | extracorporeal life | | | extracorporeal life support | extracorporeal life support | life support systems as an |
| | support systems as an | | | systems as an organ- | systems as an organ- | organ-substituting aid for |
| | organ-substituting aid for | | | substituting aid for | substituting aid for | pulmonary failure |
| | pulmonary failure | | | pulmonary failure | pulmonary failure | paintonary failure |
| | Collection of data on the | | | There will be a collection | There will be a collection | There will be a collection data |
| | inflammatory response, | | | data on inflammatory | data on inflammatory | on inflammatory response, |
| 4.2 | leukocyte function, doses | 2021 | 36 | response, leukocyte function, | response, leukocyte | leukocyte function, doses of |
| | of inotropic support after | | | doses of inotropic support | function, doses of inotropic | inotropic support after |
| | implantation of | | | after implantation of | support after implantation of | implantation of extracorporeal |

| | extracorporeal life | | | extracorporeal life support | extracorporeal life support | life support systems as an |
|---|---|---|---|---|---|---|
| | support systems as an | | | systems as an organ- | systems as an organ- | organ-substituting aid for |
| | organ-substituting aid for | | | substituting aid for | substituting aid for | pulmonary failure |
| | pulmonary failure | | | pulmonary failure | pulmonary failure | |
| | Long-term results | | | Long-term results will be | Long-term results will be | Long-term results will be |
| | collection: length of stay | | | collected: length of stay in | collected: length of stay in | collected: length of stay in the |
| | in the intensive care unit, | | | the intensive care unit, 30 | the intensive care unit, 30 | intensive care unit, 30 day |
| | 30 day survival after | | | day survival after | day survival after | |
| 4.3 | implantation of | 2021 | 36 | implantation of | implantation of | survival after implantation of |
| | extracorporeal life | | | extracorporeal life support | extracorporeal life support | extracorporeal life support |
| | support systems as an | | | systems as an organ- | systems as an organ- | systems as an organ- |
| | organ-substituting aid for | | | substituting aid for | substituting aid for | substituting aid for pulmonary |
| | pulmonary failure | | | pulmonary failure | pulmonary failure | failure |
| | Collection of laboratory | | | There will be a collection | There will be a collection | There will be a collection |
| | and clinical data, blood | | | laboratory and clinical data, | laboratory and clinical data, | laboratory and clinical data, |
| | sampling for pro- and | | | blood sampling for pro- and | blood sampling for pro- and | blood sampling for pro- and |
| 4.4 | anti-inflammatory | 2021 | 36 | anti-inflammatory cytokines, | anti-inflammatory cytokines, | anti-inflammatory cytokines, |
| | cytokines, assessment of | | | assessment of organ | assessment of organ | assessment of organ |
| | organ dysfunction, dose | | | dysfunction, doses of | dysfunction, doses of | dysfunction, doses of |
| | of vasopressors after | | | vasopressors after | vasopressors after | vasopressors after |

| | implantation of | | | implantation of | implantation of | implantation of extracorporeal |
|---|---|---|---|---|---|---|
| | extracorporeal life | | | extracorporeal life support | extracorporeal life support | life support systems as an |
| | support systems as an | | | systems as an organ- | systems as an organ- | organ-substituting aid in heart |
| | organ-substituting aid in | | | substituting aid in heart | substituting aid in heart | failure |
| | heart failure | | | failure | failure | |
| 4.5 | Collection of data on inflammatory response, leukocyte function, doses of inotropic support after implantation of extracorporeal life support systems as an organ-substituting aid in heart failure | 2021 | 36 | There will be a collection data on inflammatory response, leukocyte function, doses of inotropic support after implantation of extracorporeal life support systems as organ-substituting benefits for heart failure | There will be a collection data on inflammatory response, leukocyte function, doses of inotropic support after implantation of extracorporeal life support systems as organ- substituting benefits for heart failure | There will be a collection data on inflammatory response, leukocyte function, doses of inotropic support after implantation of extracorporeal life support systems as organ-substituting benefits for heart failure |
| 4.6 | Long-term results collection: length of stay in the intensive care unit, 30 day survival after implantation of extracorporeal life support systems as an | 2021 | 36 | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after implantation of extracorporeal life support systems as an organ- | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after implantation of extracorporeal life support systems as an organ- | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after implantation of extracorporeal life support systems as an organ-substituting aid for |

| | organ-substituting aid for | | | substituting aid for heart | substituting aid for heart | heart failure |
|---|---|---|---|---|---|---|
| | heart failure | | | failure | failure | |
| 4.7 | Collection of laboratory and clinical data, blood sampling for pro- and anti-inflammatory cytokines, assessment of organ dysfunction, dose of vasopressors after implantation of an auxiliary device of the left ventricle and implantation of a completely artificial heart as an organ-replacing aid in case of heart failure. | 2021 | 36 | There will be a collection laboratory and clinical data, blood sampling for pro- and anti-inflammatory cytokines, assessment of organ dysfunction, dose of vasopressors after implantation of an auxiliary device of the left ventricle and implantation of a completely artificial heart as an organ-replacing aid in case of heart failure | assessment of organ dysfunction, dose of vasopressors after implantation of an auxiliary | There will be a collection laboratory and clinical data, blood sampling for pro- and anti-inflammatory cytokines, assessment of organ dysfunction, dose of vasopressors after implantation of an auxiliary device of the left ventricle and implantation of a completely artificial heart as an organ-replacing aid in case of heart failure |
| 4.8 | Data collection of inflammatory response, leukocyte function, inotropic support doses after implantation of an | 2021 | 36 | There will be a collection inflammatory response data, leukocyte function, inotropic support doses after implantation of an auxiliary | There will be a collection inflammatory response data, leukocyte function, inotropic support doses after implantation of an auxiliary | There will be a collection inflammatory response data, leukocyte function, inotropic support doses after implantation of an auxiliary |

| | auxiliary device of the | | | device of the left ventricle | device of the left ventricle | device of the left ventricle and |
|---|---|---|---|---|---|---|
| | left ventricle and | | | and implantation of a | and implantation of a | implantation of a completely |
| | implantation of a | | | completely artificial heart as | completely artificial heart as | artificial heart as an organ- |
| | completely artificial heart | | | an organ-replacing aid in | an organ-replacing aid in | replacing aid in case of heart |
| | as an organ-replacing aid | | | case of heart failure. | case of heart failure. | failure. |
| | in case of heart failure. | | | | | |
| 4.9 | Long-term data collection: length of stay in the intensive care unit, 30 day survival after implantation of an auxiliary device of the left ventricle and implantation of a completely artificial heart | 2021 | 36 | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after implantation of an auxiliary device of the left ventricle and implantation of a completely artificial heart as an organ-replacing aid in | and implantation of a | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after implantation of an auxiliary device of the left ventricle and implantation of a completely artificial heart as an organ-replacing aid in case of heart |
| | as an organ-replacing aid in case of heart failure. | | | case of heart failure. | case of heart failure. | failure. |
| 4.10 | Collection of laboratory | 2021 | 36 | There will be a collection | There will be a collection | There will be a collection |
| | and clinical data, blood | | | laboratory and clinical data, | laboratory and clinical data, | laboratory and clinical data, |
| | sampling for pro- and | | | blood sampling for pro- and | blood sampling for pro- and | blood sampling for pro- and |
| | anti-inflammatory | | | anti-inflammatory cytokines, | anti-inflammatory cytokines, | anti-inflammatory cytokines, |

| | cytokines, assessment of | | | assessment of organ | assessment of organ | assessment of organ |
|---|---|---|---|---|---|---|
| | organ dysfunction, dose | | | dysfunction, dose of | dysfunction, dose of | dysfunction, dose of |
| | of vasopressors during | | | vasopressors after | vasopressors after | vasopressors after |
| | operations with | | | reconstruction of the aortic | reconstruction of the aortic | reconstruction of the aortic |
| | prolonged artificial | | | arch with long-term artificial | arch with long-term artificial | arch with long-term artificial |
| | circulation, hypothermia | | | circulation and hypothermia, | circulation and hypothermia, | circulation and hypothermia, |
| | and circulatory arrest, as | | | as an organ-replacing aid | as an organ-replacing aid | as an organ-replacing aid |
| | an organ-substituting aid | | | | | |
| 4.11 | Collection of data on inflammatory response, leukocyte function, inotropic support doses during operations with prolonged artificial circulation, hypothermia and circulatory arrest, as an organ-substituting aid | 2021 | 36 | There will be a collection inflammatory response data, leukocyte function, inotropic support doses after reconstruction of the aortic arch with long-term artificial circulation and hypothermia, as an organ-replacing aid | leukocyte function, inotropic support doses after reconstruction of the aortic arch with long-term artificial | support doses after reconstruction of the aortic arch with long-term artificial |
| 4.12 | Long-term data collection: length of stay | 2021 | 36 | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after | There will be a collection long-term results: length of stay in the intensive care unit, 30 day survival after |

| | operations with long-term | | | reconstruction of the aortic | reconstruction of the aortic | reconstruction of the aortic |
|---|---|---|---|---|---|---|
| | artificial circulation, | | | arch with long-term artificial | arch with long-term artificial | arch with long-term artificial |
| | hypothermia and | | | circulation and hypothermia, | circulation and hypothermia, | circulation and hypothermia, |
| | circulatory arrest, as an | | | as an organ-replacing aid | as an organ-replacing aid | as an organ-replacing aid |
| | organ-substituting aid | | | | | |
| | Analysis of clinical and | | | | An analysis of clinical and | An analysis of clinical and |
| | laboratory data on the | | | | laboratory data on the | laboratory data on the |
| 5 | restoration of organ | 2022 | 24 | | restoration of organ function | restoration of organ function |
| | function using innovative | | | | will be carried out using | will be carried out using |
| | technologies | | | | innovative technologies | innovative technologies |
| | Statistical processing and | | | | Statistical processing of the | Statistical processing of the |
| 6 | analysis of the obtained | 2022 | 24 | | obtained research results | obtained research results will |
| | data | | | | will be carried out | be carried out |
| | Determination of an | | | | | An effective method will be |
| | effective method of | | | | | determined of the treatment of |
| 7 | treating heart and | 2023 | 12 | | | heart and pulmonary failure |
| | pulmonary failure using | | | | | using organ replacement |
| | organ replacement | | | | | technologies |
| | technologies. | | | | | Comologics |
| 8 | Development of | 2022 | 24 | | Innovative methods of | Innovative methods of |
| | innovative methods of | 2022 | | | treating patients using | treating patients using organ- |

| | treating patients using | | | | organ-replacing technologies | replacing technologies will be |
|---|---|---|---|---|---|---|
| | organ-replacing | | | | will be developed | developed |
| | technologies | | | | | |
| 9 | Development of practical protocols for the restoration of organ function | 2022 | 24 | | Practical protocols to restore organ function will be developed | Practical protocols to restore organ function will be developed |
| 10 | Implementation of patient treatment protocols using organ-replacing technologies | 2023 | 12 | | | Patient treatment protocols using organ-replacing technologies will be introduced |
| 11 | Writing and submission of interim and final reports | 2021 | 36 | Interim report will be prepared | Interim report will be prepared | Final report will be prepared |
| 12 | Preparation of publications, reports | 2022 | 24 | | Publications will be prepared | Publications will be prepared |

# 9. Expected results of the program.

#### **Direct results:**

The obtained results of the study will form the basis for practical protocols for the use of extracorporeal life support systems, operations for the implantation of left ventricular assistive devices and a completely artificial heart.

The obtained protocols will be implemented in the treatment of patients using organreplacing technologies and will be documented.

As part of the study, innovative methods of treating patients using organ-replacing technologies will be developed:

- with the implantation of a completely artificial heart, as an organ-replacing aid, in case of heart failure;
- with implantation of an auxiliary device of the left ventricle, as an organ-replacing aid, in case of heart failure;
- when using extracorporeal life support systems in the treatment of pulmonary and / or heart failure.

The developed methods will be used as new standards and recommendations for the treatment of heart and pulmonary failure.

The developed recommendations will form the basis for a number of educational events within the framework of the ECMO School with the involvement of specialists from all regions of the country.

Will be published at least 2 (two) articles and (or) reviews in peer-reviewed scientific journals in the scientific direction of the program included in the 1 (first), 2 (second) or 3 (third) quartiles in the Web of Science database and (or) having a percentile CiteScore in the Scopus database is at least 50 (fifty).

The results of the study can help to reduce the rate of postoperative mortality in critically ill patients with pulmonary and / or heart failure by 30%.

To popularize science, a separate website will be created, which will provide complete information on the progress of the program. For each scientific publication within the framework of the program, information will be published on the website and / or in social networks.

#### **End results:**

In general, the expected efficiency and effectiveness of the proposed project will make a significant contribution to the development of the health care system in Kazakhstan, namely, to improve organ recovery, reduce postoperative complications, reduce postoperative mortality and improve the quality of life of patients.

The data obtained on the treatment of patients with heart and pulmonary failure through the use of innovative technologies will provide the necessary information to improve the quality of tertiary medical care and the quality of life of patients in Kazakhstan and around the world.

This project is aimed at achieving the indicators of the State Program for Healthcare Development 2020-2025. An increase in the average life expectancy of population up to 75 years and a decrease in the risk of premature mortality from 30 to 70 years from cardiovascular diseases.

In addition, the results will lead to modernization and an increase in the share of innovative organ-replacing technologies in the health care system.

# 10. Библиография

- 1. Starling R.C. Improved quantity and quality of life: A winning combination to treat advanced heart failure. J Am Coll Cardiol 2010;55:1835–1836.
- 2. Maciver J, Ross HJ. Quality of life and left ventricular assist device support. Circulation 2012;126:866–874.
- 3. Piergiorgio Tozzi, Roger Hullin. Mechanical circulatory support for destination therapy. Swiss Med Wkly. 2016;146:w14267.
- 4. Summer Paolone, BS, MSN, RN1. Extracorporeal Membrane Oxygenation (ECMO) for Lung Injury in Severe Acute Respiratory Distress Syndrome (ARDS): Review of the Literature. Clinical Nursing Research 2017, Vol. 26(6) 747–762
- 5. Darryl Abrams, A. Reshad Garan, Akram Abdelbary et al. Position paper for the organization of ECMO programs for cardiac failure in adults. Intensive Care Med https://doi.org/10.1007/s00134-018-5064-5.
- 6. Hunt SA. Taking heart: Cardiac transplantation past, present, and future. N Engle J Med 2006; 355: 231–35
- 7. Hunt SA, Haddad F. The changing face of heart transplantation. J Am CollCardiol 2008; 52: 587–98.

- 8. Lund LH, Edwards LB, Kucheryavaya AY, et al. The Registry of the International Society for Heart and Lung Transplantation: thirty-firstofficial adult heart transplant report-2014; focus theme: retransplantation. J Heart Lung Transplant 2014; 33: 996–1008.
- 9. Elliott MJ. Ultrafiltration and modified ultrafiltration in pedi¬atric open heart operations. Ann Thorac Surg. 1993;56(6):1518–22.6. A.M.C. Sogayar, F.R. Machado, A. Rea-Neto, A. Dornas, C.M.C. Grion, S.M.A. Lobo, et al. A multicenter, prospective study to evaluate costs of septic patients in Brazilian intensive care units Pharmacoeconomics, 26 (2008), pp. 425-434, 10.2165/00019053-200826050-00006
- 10. C. Adrie, C. Alberti, C. Chaix-Couturier, É. Azoulay, A. De Lassence, Y. Cohen, et al. Epidemiology and economic evaluation of severe sepsis in France: Age, severity, infection site, and place of acquisition (community, hospital, or intensive care unit) as determinants of workload and cost J Crit Care, 20 (2005), pp. 46-58, 10.1016/j.jcrc.2004.10.005
- 11. B. Khwannimit, R. Bhurayanontachai. The direct costs of intensive care management and risk factors for financial burden of patients with severe sepsis and septic shock J Crit Care, 30 (2015), pp. 929-934, 10.1016/j.jcrc.2015.05.011
- 12. K.N. Iskander, M.F. Osuchowski, D.J. Stearns-Kurosawa, S. Kurosawa, D. Stepien, C.Valentine, et al. Sepsis: multiple abnormalities, heterogeneous responses, and evolving understanding Physiol Rev, 93 (2013), pp. 1247-1288, 10.1152/physrev.00037.2012
- 13. A. Kwan, M. Hubank, A. Rashid, N. Klein, M.J. Peters, Transcriptional instability during evolving sepsis may limit biomarker based risk stratification PLoS One, 8 (2013), pp. 1-8, 10.1371/journal.pone.0060501
- 14. S. Akira, S. Uematsu, O. Takeuchi Pathogen recognition and innate immunity Cell, 124 (2006), pp. 783-801, 10.1016/j.cell.2006.02.015
- 15. R.S. Hotchkiss, G. Monneret, D. Payen Sepsis-induced immunosuppression: From cellular dysfunctions to immunotherapy Nat Rev Immunol, 13 (2013), pp. 862-874, 10.1038/nri3552
- 16. F. Venet, A.C. Lukaszewicz, D. Payen, R. Hotchkiss, G. Monneret Monitoring the immune response in sepsis: A rational approach to administration of immune adjuvant therapies. Curr Opin Immunol, 25 (2013), pp. 477-483, 10.1016/j.coi.2013.05.006
- 17. I. László, D. Trásy, Z. Molnár, J. FazakasSepsis: from pathophysiology to individualized patient care J Immunol Res, 2015 (2015), 10.1155/2015/510436
- 18. D.N. Cruz, M. Antonelli, R. Fumagalli, F. Foltran, N. Brienza, A. Donati, et al. Early use

- of polymyxin B hemoperfusion in abdominal septic shock, JAMA, 301 (2009), p. 2445, 10.1001/jama.2009.856
- 19. K.G. Kreymann, G. De Heer, A. Nierhaus, S. KlugeUse of polyclonal immunoglobulins as adjunctive therapy for sepsis or septic shock, Crit Care Med, 35 (2007), pp. 2677-2685, 10.1097/01.CCM.0000295263.12774.97
- R. Bellomo, I. Baldwin, C. RoncoExtracorporeal blood purification therapy for sepsis and systemic inflammation: its biological rationale, Contrib Nephrol, 132 (2001), pp. 367-374, 10.1159/000060105
- 21. Cytokine adsorber ents. The Adsorber n.d. http://Cytokine adsorber -therapy.com/the-adsorber (accessed March 5, 2018).
- R. Namas, R. Namas Hemoadsorption Reprograms Inflammation in Experimental Gramnegative Septic Peritonitis: Insights from In Vivo and In Silico Studies Mol Med, 18 (2012), p. 1, 10.2119/molmed.2012.00106
- 23. Z.Y. Peng, M.J. Carter, J.A. Kellum Effects of hemoadsorption on cytokine removal and short-term survival in septic rats, Crit Care Med, 36 (2008), pp. 1573-1577, 10.3174/ajnr.A1256
- 24. Z.Y. Peng, H.Z. Wang, M.J. Carter, M.V. Dileo, J.V. Bishop, F.H. Zhou, et al. Acute removal of common sepsis mediators does not explain the effects of extracorporeal blood purification in experimental sepsis Kidney Int, 81 (2012), pp. 363-369, 10.1038/ki.2011.320
- 25. J.A. Kellum, R. Venkataraman, D. Powner, M. Elder, G. Hergenroeder, M. CarterFeasibility study of cytokine removal by hemoabsortion in brain-dead humans, Crit Care Med, 36 (2008), pp. 268-272, 10.1097/01.CCM.0000291646.34815.BB
- 26. S. Friesecke, K. Träger, G.A. Schittek, Z. Molnar, F. Bach, K. Kogelmann, et al.International registry on the use of Cytokine adsorber ® adsorber in ICU patients: Study protocol and preliminary results, Medizinische Klin Intensivmed Und Notfallmedizin, 2017 (2017), 10.1007/s00063-017-0342-5
- 27. A.Rhodes, L.E. Evans, W. Alhazzani, M.M. Levy, M. Antonelli, R. Ferrer, et al. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock vol. 43, Springer, Berlin Heidelberg (2016, 2017), 10.1007/s00134-017-4683-6
- 28. R. Moreno, J.L. Vincent, R. Matos, A. Mendonça, F. Cantraine, L. Thijs, et al. The use of maximum SOFA score to quantify organ dysfunction/failure in intensive care. Results of a prospective, multicenter study, Intensive Care Med, 25 (1999), pp. 686-696,

## 10.1007/s001340050931

- 29. H. Hetz, R. Berger, P. Recknagel, H. SteltzerSeptic shock secondary to β-hemolytic streptococcus-induced necrotizing fasciitis treated with a novel cytokine adsorption therapy Int J Artif Organs, 37 (2014), pp. 422-426, 10.5301/ijao.5000315
- 30. K. Kogelmann, D. Jarczak, M. Scheller, M. DrünerHemoadsorption byCytokine adsorber in septic patients: A case series, Crit Care, 21 (2017), pp. 1-10, 10.1186/s13054-017-1662-9
- 31. G.W. van der Linde, A.F. Grootendorst, First case of toxic shock treated with haemoadsorption by Cytokine adsorber ® in the Netherlands, Netherlands J Crit Care, 24 (2016), pp. 27-29
- 32. S. David, K. Thamm, B.M.W. Schmidt, C.S. Falk, J.T. Kielste in Effect of extracorporeal cytokine removal on vascular barrier function in a septic shock patient, J Intensive Care, 5 (2017), pp. 1-5, 10.1186/s40560-017-0208-1
- 33. E. Nemeth, E. Kovacs, K. Racz, A. Soltesz, S. Szigeti, N. Kiss, et al., Impact of intraoperative cytokine adsorption on outcome of patients undergoing orthotropic heart transplantation an observational study, Clin Transplant (2018), 10.1111/ctr.13211
- 34. D. Trásy, K. Tánczos, M. Németh, P. Hankovszky, A. Lovas, A. Mikor, et al.Early procalci-tonin kinetics and appropriateness of empirical antimicrobial therapy in critically ill pa-tients. A prospective observational study, J Crit Care, 34 (2016), pp. 50-55, 10.1016/j.jcrc.2016.04.007
- 35. N. Öveges, I. László, M. Forgács, T. Kiss, P. Hankovszky, P. Palágyi, et al., Procalcitonin elimination during cytokine adsorption therapy in septic shock: a spin-off study of the ACESS trial Crit Care, 21 (2017), p. 383, 10.1186/s13054-017-1629-x
- 36. S. Riedel Procalcitonin and the role of biomarkers in the diagnosis and management of sepsis Diagn Microbiol Infect Dis, 73 (2012), pp. 221-227, 10.1016/j.diagmicrobio.2012.05.002
- 37. E.S. Nylen, K.T. Whang, R.H. Snider, P.M. Steinwald, J.C. White, K.L. Becker, Mortality is increased by procalcitonin and decreased by an antiserum reactive to procalcitonin in experimental sepsis, Crit Care Med, 26 (1998), pp. 1001-1006, 10.1097/00003246-199806000-00015
- 38. D. Schädler, C. Pausch, D. Heise, A. Meier-Hellmann, J. Brederlau, N. Weiler, et al. The ef-fect of a novel extracorporeal cytokine hemoadsorption device on IL-6 elimination in septic patients: A randomized controlled trial, PLoS One, 12 (2017), pp. 1-19, 10.1371/journal.pone.0187015

- 39. D. Trásy, Z. MolnárProcalcitonin assisted antibiotic strategy in sepsis, EJIFCC, 28 (2017),pp.104-11, <a href="https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5460008/pdf/ejifcc-28-104.pdf">https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5460008/pdf/ejifcc-28-104.pdf</a>
- 40. K. Tschaikowsky, S. Sägner, N. Lehnert, M. Kaul, J. Ritter Endothelin in septic patients: effects on cardiovascular and renal function and its relationship to proinflammatory cytokines, Crit Care Med, 28 (2000), pp. 1854-1860, 10.1097/00003246-200006000-00028
- 41. Benjamin E. J. et al. Heart disease and stroke statistics—2018 update: a report from the American Heart Association //Circulation. − 2018. − T. 137. − №. 12. − C. e67-e492.
- 42. Rodriguez L. E. et al. Ventricular assist devices (VAD) therapy: New technology, new hope? /Methodist DeBakey cardiovascular journal. − 2013. − T. 9. − №. 1. − C. 32.
- 43. Lietz K. et al. Outcomes of left ventricular assist device implantation as destination therapy in the post-REMATCH era: implications for patient selection //Circulation. − 2007. T. 116. № 5. C. 497-505.
- 44. Feldman D. et al. The 2013 International Society for Heart and Lung Transplantation Guidelines for mechanical circulatory support: executive summary //The Journal of Heart and Lung Transplantation. − 2013. − T. 32. − №. 2. − C. 157-187.
- 45. Hetzer R., Walter E. M. D. Trends and outcomes in heart transplantation: the Berlin experience //HSR proceedings in intensive care & cardiovascular anesthesia. 2013. T. 5. №. 2. C. 76.
- 46. Hunt S. A. Taking heart-cardiac transplantation past, present, and future //The New England journal of medicine. 2006. T. 355. № 3. C. 231.
- 47. Hunt S. A., Haddad F. The changing face of heart transplantation //Journal of the American College of Cardiology. −2008. − T. 52. − № 8. − C. 587-598.
- 48. Chen Y. F. et al. Effect of leukocyte depletion on endothelial cell activation and transendothelial migration of leukocytes during cardiopulmonary bypass //The Annals of thoracic surgery. − 2004. − T. 78. − №. 2. − C. 634-642.